CLINICAL TRIAL: NCT03975426
Title: The Use of Absorbable Screws to Treat Children and Adolescents With Anterior-Superior Iliac Spine Avulsion Fractures
Brief Title: Absorbable Screws to Treat Anterior-Superior Iliac Spine Avulsion Fractures
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yuxi Su, Vice-Dean of the Pediatric orthopedic, Children's Hospital of Chongqing Medical University
Other Study IDs: CHCMU-Yuxisu002
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Fractures, Bone; Pediatrics
MeSH Terms: conditions — Fractures, Bone | interventions — Open Fracture Reduction; Fracture Fixation, Internal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- conservative group: received conservative therapy involving bed rest with the affected lower extremity positioned with the hip and knee in flexion to ensure minimal tension of the muscles attached to the ASIS avulsion fracture.
- absorbable screws: received open reduction and internal fixation with fixation by absorbable screws.
  Interventions: Procedure: open reduction and internal fixation with fixation by absorbable screws

INTERVENTIONS:
Procedure: open reduction and internal fixation with fixation by absorbable screws — Group A received conservative therapy involving bed rest with the affected lower extremity positioned with the hip and knee in flexion to ensure minimal tension of the muscles attached to the ASIS avulsion fracture. Group B received open reduction and internal fixation with fixation by absorbable screws.
  Groups: absorbable screws

SUMMARY:
There is some debate over the best treatment for anterior-superior iliac spine (ASIS) avulsion fractures although conservative treatment can be applied when there are no neurological symptoms. Open reduction and internal fixation can be performed for dislocations exceeding 1.5 cm, or in patients requiring a short period of convalescence, although a second operation is subsequently required to extract osteosynthetic material. In this paper, we introduce the use of absorbable screws as a new fixation material for the second round of surgery.

DETAILED DESCRIPTION:
To investigate the feasibility of absorbable screws as a new fixation material for the treatment of ASIS avulsion fractures in children and adolescents.The investigator plan to retrospectively analyzed 59 patients diagnosed with ASIS avulsion fractures in our hospital between Jan 2009 and Dec 2016. These patients were divided into two groups: group A (conservative group) and group B (absorbable screws). Group A received conservative therapy involving bed rest with the affected lower extremity positioned with the hip and knee in flexion to ensure minimal tension of the muscles attached to the ASIS avulsion fracture. Group B received open reduction and internal fixation with fixation by absorbable screws. Six weeks and three months after treatment, all patients were assessed for range of motion (ROM) and by X-ray as they returned to activity. One week after treatment, the American Academy of Orthopaedic Surgeons (AAOS) lower limb and hip score was used to evaluate hip function; the same scores were also determined during follow-up at 1, 3, 6 and 12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* avulsion fracture of the ASIS
* new fractures

Exclusion Criteria:

* old avulsion fractures
* delayed fractures
* multiple fractures.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study was a retrospective review of one center's experience of treating avulsion fractures of the ASIS in children and adolescents. All patients were evaluated and treated in the same hospital.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
American Academy of Othopaedic Surgeons lower limb and hip scores | 6th month
  Stiffness of the Hip 0-5 scores, higher values represent a better outcome
American Academy of Othopaedic Surgeons lower limb and hip scores | 6th month
  swelling of the Hip 0-5 scores,higher values represent a better or worse outcome
American Academy of Othopaedic Surgeons lower limb and hip scores | 6th month
  Walking 0-5 scores ,higher values represent a better or worse outcome
American Academy of Othopaedic Surgeons lower limb and hip scores | 6th month
  Going up and goingdown stairs 0-5 ,higher values represent a better or worse outcome
American Academy of Othopaedic Surgeons lower limb and hip scores | 6th month
  bed rest 0-5 scores,higher values represent a better or worse outcome
American Academy of Othopaedic Surgeons lower limb and hip scores | 6th month
  Moving 0-5 scores,higher values represent a better or worse outcome
American Academy of Othopaedic Surgeons lower limb and hip scores | 6th month
  wear socks wear socks Wearing socks 0-5 scores,higher values represent a better or worse outcome

IPD SHARING:
Plan to Share IPD: No